CLINICAL TRIAL: NCT06149078
Title: The Relationship of Serum Uric Acid With Severity of Knee Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Saber, resident at Physical Medicine , Rheumatology and rehabilitation department, Sohag University
Other Study IDs: Soh-Med-23-11-10MS
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: hyperurecemic
  Interventions: Diagnostic Test: serum uric acid
- control group: normal
  Interventions: Diagnostic Test: serum uric acid

INTERVENTIONS:
Diagnostic Test: serum uric acid — to detect the relaton ship of serum uric acid with sevwrity of knee osteoarthritis

SUMMARY:
Osteoarthritis (OA) is the most prevalent form of arthritis. Its pathogenesis remains poorly understood. Though historically regarded as a disease of mechanical degeneration, it is now appreciated that inflammation plays an important role in OA pathogenesis (Krasnokutsky et al., 2017). The hallmark of OA is the degradation and loss of articular cartilage, although most tissues of the joint become affected, such as bone, synovium, ligaments, menisci (knee), labrum (hip), periarticular fat, and muscle (Englund, 2023).It is believed that there is a pathological link between hyperuricemia and OA Therefore, we conducted a cross-sectional study to evaluate an association between elevated SUA and radiographic OA of the knee) Bipan Shrestha, 2019 (.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (Age>18 years) with a complaint of knee pain.

Exclusion Criteria:

* 1.Any patient with a history of trauma to the knee. 2 Any patient with knee complaints as a part of autoimmune connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Adult patient (Age>18 years) with a complaint of knee pain.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
percentage of serum uric acid | 6 months
  detect the relationship of serum uric acid with severity of knee osteoarthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Englund M. Osteoarthritis, part of life or a curable disease? A bird's-eye view. J Intern Med. 2023 Jun;293(6):681-693. doi: 10.1111/joim.13634. Epub 2023 Apr 2. PMID 37004213
- [Background] Krasnokutsky S, Oshinsky C, Attur M, Ma S, Zhou H, Zheng F, Chen M, Patel J, Samuels J, Pike VC, Regatte R, Bencardino J, Rybak L, Abramson S, Pillinger MH. Serum Urate Levels Predict Joint Space Narrowing in Non-Gout Patients With Medial Knee Osteoarthritis. Arthritis Rheumatol. 2017 Jun;69(6):1213-1220. doi: 10.1002/art.40069. Epub 2017 Apr 28. PMID 28217895
- [Background] Park D, Park YM, Ko SH, Hyun KS, Choi YH, Min DU, Han K, Koh HS. Association of general and central obesity, and their changes with risk of knee osteoarthritis: a nationwide population-based cohort study. Sci Rep. 2023 Mar 7;13(1):3796. doi: 10.1038/s41598-023-30727-4. PMID 36882508